CLINICAL TRIAL: NCT03773913
Title: Integrated Community Based Health Systems Strengthening in Northern Togo: A Preliminary Mixed-Methods Study in Kozah District
Brief Title: Integrated Community Based Health Systems Strengthening Preliminary Study in Kozah Togo
Acronym: ICBHSS-Kozah
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Integrate Health (Other)
Collaborators: Ministère de la Santé et de l'Hygiène Publique, Togo (Unknown); Université de Lomé, Faculté des Sciences de la Santé, Togo (Unknown); Albert Einstein College of Medicine (Other); Montefiore Medical Center (Other); City University of New York, School of Public Health (Other)
Responsible Party: Sponsor
Other Study IDs: ICBHSS Kozah
Record Dates: First submitted 2018-11-30; First posted 2018-12-12 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Maternal-Child Health Services; Health Service Utilization
Keywords: Child Mortality; Reproductive, Maternal, Newborn, and Child Health; Community Health Workers; Implementation Research; Preliminary Research; Health Systems Strengthening
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Four facilities in Kozah District: Baseline estimated population of 33,412 served by four public sector facilities in Kozah District.
  Interventions: Other: ICBHSS model

INTERVENTIONS:
Other: ICBHSS model — Bundle of evidence-based interventions that include the following 5 components:
  1. Community engagement meetings and feedback;
  2. Elimination of public sector facility user fees for children under five and pregnant women;
  3. Pro-active community based IMCI using trained, equipped, supervised, and salaried Community Health Workers (CHWs) with additional services including linkage to family planning and counseling, HIV testing & referrals;
  4. Clinical mentoring and enhanced supervision by a trained peer coach at public sector facilities;
  5. Basic infrastructure improvements and supply chain management training of pharmacy managers

SUMMARY:
This preliminary study aims to inform the design and delivery of the integrated facility and community-based health systems strengthening (ICBHSS) model in four Kozah District health facilities over a period of 48 months. Specific aims include: (1) Assess maternal and child health outcomes and health service utilization rates in the 4 ICBHSS model intervention sites catchment areas; (2) Identify barriers to and facilitators of access and quality services related to ICBHSS model; and (3) Assess changes in health care services coverage, effectiveness, and adoption of ICBHSS model.

DETAILED DESCRIPTION:
Intervention: The investigators have adapted an integrated facility and community-based health systems strengthening (ICBHSS) model to improve primary healthcare services in Togo. The ICBHSS model includes a bundle of evidence based interventions including (1) community engagement meetings and feedback; (2) the elimination of facility user fees for children under five and pregnant women; (3) pro-active community based IMCI using Community Health Workers (CHWs) with additional services including linkage to family planning and counseling, HIV testing & referrals; (4) clinical mentoring and enhanced supervision at public sector facilities; and (5) improved supply chain management and facility structures.

Study: The investigators will conduct a mixed methods assessment, using the RE-AIM framework to evaluate the impact and implementation of the ICBHSS initiative in Kozah district. It will include: (1) a repeated cross-sectional study to obtain annual coverage, effectiveness, and adoption metrics using a population-based household survey as well as (2) qualitative key informant interviews and focus group discussions conducted at 12 months for each intervention health facility. The primary outcome will be under 5 year old mortality rate, with secondary outcomes including under-one mortality rate, maternal mortality rate, as well as maternal and child health service utilization.

ELIGIBILITY:
Inclusion Criteria:

* Female of reproductive age (aged 15-49 years)
* Individuals aged 15-17 years will only be included if they have children and/or are pregnant
* Lives in selected household within study catchment area
* Informed consent is obtained for participants 18-49
* Waiver of parental permission is obtained for 15-17 year-old participants

Exclusion Criteria:

-

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Females of reproductive age (aged 15-49 years) who reside in a selected household within the study catchment area.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Under-five year old mortality rate, annual | 72 months
  The under-five mortality rate (expressed as a rate per 1,000 live births) is the probability of a child dying in a specified year between birth and 5 years of age.

SECONDARY OUTCOMES:
Under-one year old mortality rate, annual | 72 months
  The under-one mortality rate (expressed as a rate per 1,000 live births) is the probability of a child dying in a specified year between birth and 1 year of age.
Maternal mortality rate, annual | 72 months
  The maternal mortality rate (expressed as a rate per 100,000 live births) is the probability of a mother dying in a specified year within 42 days of pregnancy termination.
Annual proportion of children under age five reported to be febrile in the prior two weeks who received an effective antimalarial treatment within 24 hours of symptom onset. | 72 months
  The number of febrile children under-five who received an effective antimalarial treatment within 24 hours of symptom onset out of the total number of children under age five reported to be febrile in the prior two weeks.
Annual proportion of children under age five reported to have a cough in the prior two weeks who received an effective pneumonia treatment within 24 hours of symptom onset. | 72 months
  The number of children under-five who received an effective pneumonia treatment within 24 hours of symptom onset out of the total number of children under age five reported to have a cough in the prior two weeks.
Annual proportion of children under age five reported to have diarrhea in the prior two weeks who received an effective treatment for diarrheal disease within 24 hours of symptom onset. | 72 months
  The number of children under-five who received an effective treatment for diarrheal disease within 24 hours of symptom onset out of the total number of children under age five reported to have diarrhea in the prior two weeks.
Maternal facility based birth delivery incidence rate, annual | 72 months
  The proportion of women reported to have delivered in a health facility.
Protocol Adherence by IH community health workers in iCCM and maternal consultations | 72 months
  The average adherence by IH community health workers to evidence-based protocols for iCCM and maternal consultations as measured by CHW supervisor check-list.
Protocol adherence by clinical staff at IH intervention facilities in iCCM and maternal consultations | 72 months
  The average adherence by public sector clinical staff at IH intervention sites to evidence-based protocols for iCCM and maternal consultations as measured by IH clinical mentor supervision check-list.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin P Fiori Jr., MD MPH, Principal Investigator — Integrate Health; Albert Einstein School of Medicine; Molly E Lauria, MPH, Study Director — Integrate Health
Locations (1):
- Integrate Health, Kara, Togo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fiori K, Schechter J, Dey M, Braganza S, Rhatigan J, Houndenou S, Gbeleou C, Palerbo E, Tchangani E, Lopez A, Bensen E, Hirschhorn LR. Closing the delivery gaps in pediatric HIV care in Togo, West Africa: using the care delivery value chain framework to direct quality improvement. AIDS Care. 2016 Mar;28 Suppl 2(sup2):29-33. doi: 10.1080/09540121.2016.1176678. PMID 27391996
- [Derived] Fiori KP, Lauria ME, Singer AW, Jones HE, Belli HM, Aylward PT, Agoro S, Gbeleou S, Sowu E, Grunitzky-Bekele M, Singham Goodwin A, Morrison M, Ekouevi DK, Hirschhorn LR. An Integrated Primary Care Initiative for Child Health in Northern Togo. Pediatrics. 2021 Sep;148(3):e2020035493. doi: 10.1542/peds.2020-035493. PMID 34452981
- [Derived] Kaplowitz ET, Fiori KP, Lauria ME, Gbeleou S, Miziou A, Sowu E, Schechter J, Jones HE. Sexual Relationship Power and Socio-demographic Factors Predicting Contraceptive Use, Antenatal Visits and Sick Child Health Service Use in Northern Togo. Matern Child Health J. 2020 Jul;24(7):845-855. doi: 10.1007/s10995-020-02948-w. PMID 32347439
- See also: Integrate Health — http://integratehealth.org/